CLINICAL TRIAL: NCT04347083
Title: A New Method to Determine Onset Point of Mechanical Stimulation Inducing Muscle Spindle-Based Stretch Reflex by Using Intramuscular Electromyography Electrodes
Brief Title: Determination of Onset Point of Mechanical Stimulation
Acronym: TrueRL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan KARACAN, Researcher and Trainer, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ISTPMR
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Reflex, Abnormal
MeSH Terms: conditions — Reflex, Abnormal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): Reflex latency will be measured in this arm
  Interventions: Diagnostic Test: Electrodiagnostic test

INTERVENTIONS:
Diagnostic Test: Electrodiagnostic test — Muscle spindle- based reflex latency will be measured

SUMMARY:
The difference between latencies of the tonic vibration reflex or T-reflex and whole body vibration-induced muscular reflex may be related to the distance between their stimulation point and the muscle spindles. Achilles tendon is mechanically stimulated by using a local vibrator to elicit the tonic vibration reflex or a reflex hammer to elicit the T-reflex. Whole body vibration, however, stimulates the soleus muscle indirectly over the heel, not directly, since whole body vibration is administered in a position that the subjects are standing on the whole body vibration platform. In other words, while the local vibrator or the hammer stimulates the Achilles tendon, whole body vibration stimulates the sole of the foot. During whole body vibration, mechanical vibration stimuli need to go a long way to reach the soleus muscle spindle. Therefore, whole body vibration-induced muscular reflex latency may be longer than tonic vibration reflex or T-reflex latency. The aim this study is to define a method for determination of onset point of mechanical stimulation inducing muscle spindle-based reflex (e.g., tonic vibration reflex, T-reflex) by using intramuscular electromyography electrodes.

DETAILED DESCRIPTION:
The aim of this study is to define a method for the determination of the onset point of mechanical stimulation inducing muscle spindle-based reflex by using Intramuscular electromyography electrodes. This research protocol has two phases: First, the method of measuring latency using MAS was described in Experiment-I. The validity of this method was then determined in Experiment II. Eight healthy volunteers will participate in experiment-I and five healthy volunteers will participate in experiment II. Two surface electromyography electrodes will be placed on the left gastrocnemius muscle belly to record spindle-based reflex response. Single motor unit electrode pairs will be then inserted between two surface electrodes into the lateral gastrocnemius muscle to record stimulus artifact caused by tapping. The Achilles tendon will be tapped 20 times at 3-5 s intervals by a reflex hammer (Achilles tapping). Participants will be then asked to stand up and stand upright on the left foot. To maintain static balance, participants will be asked to hold the handles on the wall. The left heel will be tapped 20 times at 3-5 s intervals by a hammer (Heel tapping). In experiment II, the records from multiple sites gastrocnemius lateralis and rectus femoris) will be taken to characterize how movement artifacts change based on the location of the recording electrode. Using electric signals of the switch system as the trigger and the signals recorded by intramuscular electrodes and accelerometer as the source, spike-triggered averaging was used to determine the lag time it takes for the mechanical stimulus to reach the belly of the gastrocnemius and rectus femoris muscles. Meanwhile, the internal delay time of the accelerometers (the time between the mechanical stimulus moment and the signal output moment from the accelerometer) was determined. Using electric signals of the switch system as the trigger and the signals of accelerometers as the source, spike-triggered averaging was used to determine the internal delay time of accelerometers.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* 20-45 aged
* Healthy volunteer

Exclusion Criteria:

* People with any health problems

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
muscle spindle- based reflex latency | 1 day (a single point in time)
  Duration between the onset point of mechanical stimulation and onset point of muscle spindle- based reflex latency response is defined as "muscle spindle- based reflex latency".

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan Karacan, Assoc Prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karacan I, Cidem M, Cidem M, Turker KS. Whole-body vibration induces distinct reflex patterns in human soleus muscle. J Electromyogr Kinesiol. 2017 Jun;34:93-101. doi: 10.1016/j.jelekin.2017.04.007. Epub 2017 Apr 24. PMID 28457998
- [Result] Yildirim MA, Topkara B, Aydin T, Paker N, Soy D, Coskun E, Ones K, Bardak A, Kesiktas N, Ozyurt MG, Celik B, Onder B, Kilic A, Kucuk HC, Karacan I, Turker KS. Exploring the receptor origin of vibration-induced reflexes. Spinal Cord. 2020 Jun;58(6):716-723. doi: 10.1038/s41393-020-0419-5. Epub 2020 Jan 15. PMID 31942042
- [Result] Aydin T, Kesiktas FN, Baskent A, Karan A, Karacan I, Turker KS. Cross-training effect of chronic whole-body vibration exercise: a randomized controlled study. Somatosens Mot Res. 2020 Jun;37(2):51-58. doi: 10.1080/08990220.2020.1720635. Epub 2020 Feb 5. PMID 32024411
- [Result] Cakar HI, Cidem M, Sebik O, Yilmaz G, Karamehmetoglu SS, Kara S, Karacan I, Turker KS. Whole-body vibration-induced muscular reflex: Is it a stretch-induced reflex? J Phys Ther Sci. 2015 Jul;27(7):2279-84. doi: 10.1589/jpts.27.2279. Epub 2015 Jul 22. PMID 26310784
- [Result] Karacan I, Cakar HI, Sebik O, Yilmaz G, Cidem M, Kara S, Turker KS. A new method to determine reflex latency induced by high rate stimulation of the nervous system. Front Hum Neurosci. 2014 Jul 18;8:536. doi: 10.3389/fnhum.2014.00536. eCollection 2014. PMID 25100978